CLINICAL TRIAL: NCT06395155
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Pharmacokinetic Drug-drug Interactions Between DHP2306R1 and DHP2306R2 in Healthy Adult Volunteers
Brief Title: A Phase 1 Clinical Trial DHP2306R1 and DHP2306R2 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daehwa Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2306CS-1
Record Dates: First submitted 2023-11-07; First posted 2024-05-02 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2023-10

CONDITIONS: Musculoskeletal Pain
Keywords: Phase 1; DDI; rheumatoid arthritis; degenerative arthritis; acute pain
MeSH Terms: conditions — Musculoskeletal Pain; Arthritis, Rheumatoid; Osteoarthritis; Acute Pain

STUDY DESIGN:
Intervention Model Description: Randomized, Open-label, Multiple-dose, Six-sequence, Three-period, Three-treatment, Crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence A (Experimental): DHP2306R1 100mg twice a day for 4 days, and DHP2306R1 100mg once for a day, followed by 1week of wash out period; then DHP2306R2 75mg twice a day for 4days, and DHP2306R2 75mg once for a day, followed by 1 week of wash out period; then DHP2306R1 100mg+ DHP2306R2 75mg twice a day for 4ayds and DHP2306R1 100mg+ DHP2306R2 75mg once for a day
  Interventions: Drug: DHP2306R1; Drug: DHP2306R2
- Sequence B (Experimental): DHP2306R1 100mg twice a day for 4 days, and DHP2306R1 100mg once for a day, followed by 1week of wash out period; then DHP2306R1 100mg+ DHP2306R2 75mg twice a day for 4ayds and DHP2306R1 100mg+ DHP2306R2 75mg once for a day, followed by 1 week of wash out period; then DHP2306R2 75mg twice a day for 4days, and DHP2306R2 75mg once for a day
  Interventions: Drug: DHP2306R1; Drug: DHP2306R2
- Sequence C (Experimental): DHP2306R2 75mg twice a day for 4days, and DHP2306R2 75mg once for a day, followed by 1 week of wash out period; then DHP2306R1 100mg twice a day for 4 days, and DHP2306R1 100mg once for a day, followed by 1week of wash out period; then DHP2306R1 100mg+ DHP2306R2 75mg twice a day for 4ayds and DHP2306R1 100mg+ DHP2306R2 75mg once for a day
  Interventions: Drug: DHP2306R1; Drug: DHP2306R2
- Sequence D (Experimental): DHP2306R2 75mg twice a day for 4days, and DHP2306R2 75mg once for a day, followed by 1 week of wash out period; then DHP2306R1 100mg+ DHP2306R2 75mg twice a day for 4ayds and DHP2306R1 100mg+ DHP2306R2 75mg once for a day; then DHP2306R1 100mg twice a day for 4 days, and DHP2306R1 100mg once for a day, followed by 1week of wash out period
  Interventions: Drug: DHP2306R1; Drug: DHP2306R2
- Sequence E (Experimental): DHP2306R1 100mg+ DHP2306R2 75mg twice a day for 4ayds and DHP2306R1 100mg+ DHP2306R2 75mg once for a day; then DHP2306R1 100mg twice a day for 4 days, and DHP2306R1 100mg once for a day, followed by 1week of wash out period; then DHP2306R2 75mg twice a day for 4days, and DHP2306R2 75mg once for a day, followed by 1 week of wash out period
  Interventions: Drug: DHP2306R1; Drug: DHP2306R2
- Sequence F (Experimental): DHP2306R1 100mg+ DHP2306R2 75mg twice a day for 4ayds and DHP2306R1 100mg+ DHP2306R2 75mg once for a day; then DHP2306R2 75mg twice a day for 4days, and DHP2306R2 75mg once for a day, followed by 1 week of wash out period ; then DHP2306R1 100mg twice a day for 4 days, and DHP2306R1 100mg once for a day, followed by 1week of wash out period
  Interventions: Drug: DHP2306R1; Drug: DHP2306R2

INTERVENTIONS:
Drug: DHP2306R1 — 100mg per capsule, BID
Drug: DHP2306R2 — 75mg per Tab, BID

SUMMARY:
This phase 1 study is to evaluate the safety and pharmacokinetic drug interactions of DHP2306R1 and DHP2306R2 when administered alone and in combination in healthy conditions.

Participants will be taken DHP2306R1 and DHP2306R2 alone or combination for 3 period, randomized in six-sequence.

ELIGIBILITY:
Inclusion Criteria:

* 1) Healthy adult volunteers aged 19 years or older at the time of screening
* 2) At the time of screening, those who weigh more than 50.0 kg and have a body mass index (BMI) of 18.0 kg/m2 or more and 30.0 kg/m2 or less.
* 3) Those who do not have congenital or chronic diseases requiring treatment and no pathological symptoms or findings as a result of internal medical examination
* 4) At the time of screening, those who were determined to be suitable subjects for clinical trials as a result of tests such as clinical laboratory tests, vital signs, physical examination (physical examination), and 12-lead electrocardiogram conducted according to the characteristics of the clinical trial drug.
* 5) A person who, after receiving a detailed explanation of this clinical trial and fully understanding it, voluntarily decides to participate and agrees in writing to comply with the subject compliance requirements during the clinical trial period

Exclusion Criteria:

* 1) Current or past medical history of clinically significant liver, kidney, nervous system, mental, respiratory, endocrine, blood disease, tumor, genitourinary, cardiovascular, digestive, and musculoskeletal systems, as well as the following symptoms or history. Those who have

  ① Renal impairment

  ② Liver disorder
* 2) For women, pregnant women (Urine-HCG positive) or lactating women
* 3) Persons with a history of hypersensitivity or clinically significant hypersensitivity to DHP2306R1, DHP2306R2, or components of clinical investigational drugs, aspirin, non-steroidal anti-inflammatory drugs (including COX-2 inhibitors), or sulfonamide drugs.
* 4) People with genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
* 5) Those with a history of gastrointestinal disease (Crohn's disease, ulcer, acute or chronic pancreatitis, etc.) or gastrointestinal surgery (excluding simple appendectomy or hernia surgery) that may affect the absorption of clinical trial drugs
* 6) At the time of screening, those with clinically significant findings including the following findings on 12-lead electrocardiography

  * QTc > 450 ms for men, QTc > 470 ms for women
  * PR interval > 200 ms
  * QRS duration > 120 ms
* 7) At the time of screening, a person who shows the following results in clinical laboratory tests

  * Those whose AST, ALT, ALP, γ-GT and Bilirubin total exceed twice the upper limit of the normal range in clinical laboratory tests to evaluate liver function
  * If the blood creatinine level exceeds the reference range or the eGFR calculated by CKD-EPI is less than 60 mL/min/1.73m2
  * Those whose CPK exceeds 2.5 times the upper limit of the normal range in clinical laboratory tests
* 8) If you have a history of drug abuse or test positive for drugs of abuse in a urine drug test
* 9) At the time of screening, those who showed vital signs measured in a sitting position after resting for more than 3 minutes include systolic blood pressure ≥ 150 mmHg or ≤ 90 mmHg, diastolic blood pressure ≥ 100 mmHg or ≤ 60 mmHg, and pulse ≤ 40 bpm or ≥ 100 bpm.
* 10) Persons who administered drugs that induce or inhibit drug metabolizing enzymes such as barbiturates within 1 month before the first administration date
* 11) People who eat abnormal diets that may affect the absorption, distribution, metabolism, and excretion of investigational drugs or who consume foods that may affect drug metabolism
* 12) Any prescription drugs or herbal preparations that may affect the characteristics of investigational drugs, including cyclosporine, were administered within 2 weeks before the first administration date, or any over-the-counter drugs (OTC drugs) or vitamin preparations were administered within 10 days. (However, if the drug does not affect the pharmacokinetic properties of the clinical trial drug, the applicant may participate in the clinical trial at the discretion of the investigator.)
* 13) Those who participated in and received treatment in another clinical trial within 6 months prior to the date of first administration (however, the end standard for participation in other clinical trials is based on the date of last administration, and the next day is calculated as 1 day)
* 14) Those who have donated whole blood within 2 months before the first administration date or component blood donation within 1 month, received a blood transfusion within 1 month, or cannot refrain from donating blood from the time of written consent to the time of PSV
* 15) Those who have continuously drank alcohol (exceeding 21 units/week, 1 unit=10 g=12.5 mL of pure alcohol) within 6 months before the first administration date or who are unable to abstain from drinking from the time of written consent to the time of PSV
* 16) Smokers who smoked more than 10 cigarettes on average per day within 3 months before the first administration date and those who were unable to quit smoking from 24 hours before the first administration to the time of the last blood collection in each period
* 17) Those who consumed food containing grapefruit (grapefruit) from 48 hours before the first administration until the time of PSV or who cannot refrain from consuming it
* 18) Those who consumed or were unable to refrain from consuming caffeine-containing foods (coffee, green tea, black tea, carbonated drinks, coffee milk, tonic drinks, etc.) during the period from 24 hours before the first administration in each period until the last blood collection.
* 19) Those who engaged in vigorous exercise exceeding the level of daily life during the period from 48 hours before the first administration to the time of PSV, or who cannot refrain from vigorous exercise
* 20) From the time of written consent until 2 weeks after the last date of administration of the investigational drug, even if you, your spouse, or partner are planning to become pregnant or are not planning to become pregnant, you must use reliable contraceptive methods (e.g., administration of contraceptives and implantation or intrauterine device, sterilization procedure ( Those who are not using vasectomy, tubal ligation, etc.) or barrier methods (combined use of spermicides, condoms, contraceptive diaphragms, vaginal sponges, or cervical caps))
* 21) Persons judged by the investigator to be unsuitable for participation in clinical trials due to reasons other than the above selection/exclusion criteria

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-10-26 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss of DHP2306R1 and DHP2306R2 | At baseline(Day 1 0 hours), Administration day (Day 4 to Day 5) in each period
  Systemic exposure of DHP2302R1 and DHP2302R2
Cmax of DHP2306R1 and DHP2306R2 | At baseline(Day 1 0 hours), Administration day (Day 4 to Day 5) in each period
  Plasma concentrations of DHP2306R1 and DHP2306R2

SECONDARY OUTCOMES:
AUC0-48 of DHP2306R1 and DHP2306R2 | At baseline(Day 1 0 hours), Administration day (Day 4 to Day 5) in each period
  Secondary pharmacokinetic parameters of DHP2306R1 and DHP2306R2
AUCinf of DHP2306R1 and DHP2306R2 | At baseline(Day 1 0 hours), Administration day (Day 4 to Day 5) in each period
  Secondary pharmacokinetic parameters of DHP2306R1 and DHP2306R2
Tmax of DHP2306R1 and DHP2306R2 | At baseline(Day 1 0 hours), Administration day (Day 4 to Day 5) in each period
  Secondary pharmacokinetic parameters of DHP2306R1 and DHP2306R2
t1/2 of DHP2306R1 and DHP2306R2 | At baseline(Day 1 0 hours), Administration day (Day 4 to Day 5) in each period
  Secondary pharmacokinetic parameters of DHP2306R1 and DHP2306R2
CL/F of DHP2306R1 and DHP2306R2 | At baseline(Day 1 0 hours), Administration day (Day 4 to Day 5) in each period
  Secondary pharmacokinetic parameters of DHP2306R1 and DHP2306R2
Vz/F of DHP2306R1 and DHP2306R2 | At baseline(Day 1 0 hours), Administration day (Day 4 to Day 5) in each period
  Secondary pharmacokinetic parameters of DHP2306R1 and DHP2306R2

CONTACTS AND LOCATIONS:
Overall Officials: Min Kyu Park, Principal Investigator — Chungbuk National University Hospital
Locations (1):
- Chungbuk National University Hospital, Jungbuk, South Korea